CLINICAL TRIAL: NCT01998373
Title: The Effect of Group Training on the Quality of Life and Reduction of Pain in Rheumatoid Arthritis Patients
Brief Title: Group Training and Quality of Life and Reduction of Pain in Rheumatoid Arthritis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Khazaeipour, Principal Investigator, Tehran University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 7971
Record Dates: First submitted 2013-11-18; First posted 2013-11-28 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Training Leaflet; Training Workshop
Keywords: Patient training; Rheumatoid arthritis; Quality of life
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patient training and patient without training (Experimental): Experimental group 1: patient education intervention group (PIGE) Experimental group 2: patient without intervention group (PWIG)
  Interventions: Behavioral: training leaflet and oral training
- control without education (No Intervention): this group did not receive an education

INTERVENTIONS:
Behavioral: training leaflet and oral training — The intervention consisted of training leaflet and oral training. All of the patients were new cases and were divided into 2 groups. All patients were treated with routine medication, no addition medication for two groups were done, the case group attended the workshops and were trained In addition to medical therapy, continuing education and training workshop. The result of the effect of workshop was also filling out a questionnaire before and after training. Finally, two groups with statistical analysis were compared.
  Other Names: education; training workshop
  Arms: patient training and patient without training

SUMMARY:
Abstract

Background:

It is documented that some patient education interventions, preferably with a behavioral component included, may improve pain, disability and moods Purpose of the study: the purpose of this study was to improve the quality of life and reduce pain in rheumatoid arthritis patients.

Methods:

Patients were allocated to a patient training intervention group and patient without training intervention group. Both groups received routine treatments while the patient training intervention group, in addition to the routine treatments received training booklets and participated in the training workshop. All the extracted data from the written questionnaire were collected and analyzed using SPSS software.

DETAILED DESCRIPTION:
Results:

The improvement in the signs of recovery for physical and mood symptoms in the patient training intervention group were seen (p < 0.05). The score of quality of life had significantly improved in the two groups (Mean difference was 9.31±3.03 and P<0.003). This improvement was significantly higher in the patient training intervention group (P=0.008). After adjustment for education level, the score of quality of life in patient training intervention group had a higher improvement, but the difference between the two groups was not significant (P = 0.1).

Conclusions:

This study showed the important role of training and the patients' educational level on better treatments. The appropriate training in the patient could create a change in the treatment process and has a better effect on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* The only inclusion criterion was that the patient had RA as the main disease (with the same duration and severity of disease).

Exclusion Criteria:

* Patients were excluded if they had another disease.

Ages: 34 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2006-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
The score of quality of life had significantly improved in the two groups (using questionnaire) | one year

SECONDARY OUTCOMES:
In the present study a greater percentage of patients reported less pain after intervention (using questionnaire) | one year

CONTACTS AND LOCATIONS:
Locations (1):
- the rheumatology clinic at Imam Khomeini Hospital in Tehran, Tehran, Tehran Province, Iran